CLINICAL TRIAL: NCT00129363
Title: A Multicenter, Open Label Extension Study to Evaluate the Safety of Twice Daily Oral Carvedilol in Pediatric Patients With Chronic Heart Failure
Brief Title: Study to Evaluate the Safety of Twice Daily Oral Carvedilol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shaddy, Robert, M.D. (Individual)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Robert E Shaddy, MD, The Children's Hospital of Philadelphia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB 105517-396
Record Dates: First submitted 2005-08-08; First posted 2005-08-11 (Estimated); Last update posted 2008-12-25 (Estimated); Status verified 2008-12

CONDITIONS: Congestive Heart Failure
Keywords: Adolescent; Adrenergic alpha-Antagonists/therapeutic use; Adrenergic alpha-Antagonists/pharmacokinetics; Adrenergic alpha-Antagonists/administration & dosage; Adrenergic beta-Antagonists/therapeutic use; Adrenergic beta-Antagonists/pharmacokinetics; Adrenergic beta-Antagonists/administration & dosage; Age Factors; Carbazoles/therapeutic use; Carbazoles/administration & dosage; Child; Child, Preschool; Drug Administration Schedule; Female; Heart Failure, Congestive/etiology; Heart Failure, Congestive/drug therapy; Heart Failure, Congestive/blood; Human; Infant; Infant, Newborn; Male; Natriuretic Peptide, Brain/blood; Placebos; Propanolamines/therapeutic use; Propanolamines/administration & dosage; Prospective Studies; Support, Non-U.S. Gov't; Treatment Outcome; Ventricular Dysfunction/drug therapy; Ventricular Dysfunction/complications; Ventricular Dysfunction/blood; Ventricular Function/drug effects; Ventricular Remodeling/drug effects
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction | interventions — Carvedilol

INTERVENTIONS:
Drug: Carvedilol

SUMMARY:
The objective of this study is to evaluate the long-term safety of carvedilol in pediatric patients with chronic heart failure, who completed the Pediatric Carvedilol Study 321. Carvedilol will be provided as open-label therapy for a period of at least 6 months (or until termination of the study) by SmithKline Beecham Corporation d/b/a GlaxoSmithKline (GSK) or the University Sponsor.

DETAILED DESCRIPTION:
This open-label, uncontrolled, extension study is designed to assess the long-term safety of carvedilol in pediatric patients with heart failure and includes the following phases:

1. Screening Phase (coincides with the final maintenance Month 6 Visit in the 321 study
2. Down-/Up-titration Phase
3. Maintenance Phase
4. Down-titration
5. Follow-up

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with chronic symptomatic congestive heart failure (CHF) due to systemic ventricular systolic dysfunction, who are receiving standard heart failure therapy and have successfully completed the maintenance phase of the Pediatric Carvedilol Study 321.
* Parent or guardian of patient able and willing to give written informed consent. The written assent from children > 9 years of age is also required.

Exclusion Criteria:

* A patient who, in the opinion of the investigator, would not benefit from open-label carvedilol.
* A patient who, in the opinion of the investigator, is incapable of cooperating with the requirements of this study.
* A patient treated with the following medications at the time of entry in the study:

  * Monoamine oxidase (MAO) inhibitors;
  * Calcium entry blockers;
  * α- blockers, or labetalol;
  * Disopyramide, flecainide, encainide, moricizine, propafenone;
  * Intravenous inotropes such as dobutamine or intravenous vasodilator agents such as amrinone or milrinone;
  * Intravenous CHF medications (e.g. diuretics, digoxin);
  * Beta-blockers, other than double-blind carvedilol.
* Uncorrected primary obstructive or severe regurgitative valvular disease, nondilated (restrictive) or hypertrophic cardiomyopathy, or significant systemic ventricular outflow obstruction.
* A patient with any of the following contra-indications to beta-blocker therapy:

  * Heart rate < 2nd percentile for age;
  * Unacceptable blood pressure. Sitting (supine in infants) systolic blood pressure must be > 85 mm Hg in teens; >75 mm Hg in school-aged children; and >65 mm Hg in infants;
  * Sick sinus syndrome, second or third degree atrioventricular (AV) block, unless treated with a permanent pacemaker;
  * History or current clinical evidence of moderate-to-severe obstructive pulmonary disease or reactive airway diseases (e.g., asthma) requiring therapy;
  * Unstable insulin-dependent diabetes mellitus.
* Renovascular hypertension or evidence of pulmonary hypertension (pulmonary vascular resistance index > 6 Wood units m2) unresponsive to vasodilator agents such as oxygen, nitroprusside, or nitric oxide
* A patient with any one of these general exclusion criteria:

  * Significant renal (serum creatinine > 2.0), hepatic (serum AST and/or ALT > 3 times upper limit of normal), gastrointestinal, or biliary disorders that could impair absorption, metabolism, or excretion of orally administered medications;
  * Endocrine disorders such as pheochromocytoma, active hyperthyroidism and untreated hypothyroidism;
  * Any illness other than heart failure that may limit survival within 1 year (e.g. neoplasm);
  * Girls of childbearing potential who are pregnant or sexually active and not taking adequate contraceptive precautions (e.g., intrauterine device [IUD] or oral contraceptives).
* A patient who received any investigational drug within the preceding 30 days except blinded medication in Pediatric Carvedilol Study 321. An investigational drug is defined as any agent (placebo or drug) dispensed as part of a research study.

Ages: 1 Day to 17 Years | Sex: All
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2002-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
dose tolerability
growth and development
physical exam (PE) including cardiopulmonary examination
blood pressure (BP), heart rate (HR), height (Ht) and weight [Wt] (including %)
laboratory safety assessments
pregnancy test, if applicable
an echocardiographic measurement
reporting of all adverse events [AEs] (serious and non-serious)

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Shaddy, MD, Principal Investigator — University of Utah
Locations (17):
- United States (17):
  - Mattel Children's Hospital at UCLA, Los Angeles, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Colorado, Denver, Colorado
  - University of Miami, Miami, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - Children's Hospital, Boston, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Columbia University, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Childrens Hospital and Regional Medical Center, Seattle, Washington